CLINICAL TRIAL: NCT03260361
Title: Combined Therapy of Hypnosis Kinesitherapy and MEOPA in Patients With Regional Painful Syndrome Complex
Brief Title: Hypnosis and MEOPA in Regional Painful Syndrome Complex
Acronym: ProHKM-SDRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/16/8235
Record Dates: First submitted 2017-01-24; First posted 2017-08-24 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Algodystrophy of Hand
MeSH Terms: interventions — Hypnosis; Meopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnosis Kinesitherapy and MEOPA (Experimental): combined therapy of Hypnosis Kinesitherapy and MEOPA (HKM)
  Interventions: Other: Hypnosis, kinesitherapy, MEOPA
- usual practice (Other): physiopathology and treatments
  Interventions: Other: Usual practice

INTERVENTIONS:
Other: Hypnosis, kinesitherapy, MEOPA — classical intervention
  Other Names: Hypnosis Kinesitherapy and MEOPA (HKM)
  Arms: Hypnosis Kinesitherapy and MEOPA
Other: Usual practice — Usual practice with treatments and physio
  Arms: usual practice

SUMMARY:
Relation between hypnosis and MEOPA on algodystrophy.

ELIGIBILITY:
Inclusion Criteria:

* Regional Painful Syndrome Complex

Exclusion Criteria:

* deaf people

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Pain intensity measure using visual analogical ladder (EVA) | 3 weeks
  pain intensity is determined by patient himself on a visual analogical ladder created by Huskisson

SECONDARY OUTCOMES:
QDSA ( Saint Antoine Pain Questions) | 3 weeks
  description of the type of pain
SF36 (Short Form (36) Health Survey) | 3 weeks
  quality of life appreciation
HADs | 3 weeks
  Hospital Anxiety and Depression Scale

CONTACTS AND LOCATIONS:
Overall Officials: Martine QUINTARD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - Croix du Sud, Quint-Fonsegrives
  - University Hospital of Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oerlemans HM, Oostendorp RA, de Boo T, Perez RS, Goris RJ. Signs and symptoms in complex regional pain syndrome type I/reflex sympathetic dystrophy: judgment of the physician versus objective measurement. Clin J Pain. 1999 Sep;15(3):224-32. doi: 10.1097/00002508-199909000-00010. PMID 10524476